CLINICAL TRIAL: NCT03939338
Title: Combination With Regulatory T Cell Levels and Cardiac Magnetic Resonance Imaging (CMR) to Assess the Severity and Prognosis of Reperfusion Injury After Primary PCI in STEMI Patients (TregCMRRS)
Brief Title: Combination With Treg Levels and CMR to Assess the Severity and Prognosis of Reperfusion Injury After PPCI in STEMI Patients
Acronym: TregCMRRS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hongwei Li, MD, Prof., Beijing Friendship Hospital
Other Study IDs: BFH-Treg and CMR
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; Reperfusion Injury, Myocardial
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Reperfusion Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participates
  Interventions: Other: Treg levels and CMR results

INTERVENTIONS:
Other: Treg levels and CMR results — This is an observational study. Exposure: Different Treg levels and CMR results.

SUMMARY:
This study aims to determine whether combination with regulatory T cell (Treg) levels and cardiac magnetic resonance imaging (CMR) are predictive of the severity of reperfusion injury following myocardial infarction and the prognosis in STEMI patients receiving primary percutaneous coronary intervention (PPCI).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed STEMI diagnosis
* Undergoing primary percutaneous coronary intervention (presenting <12 hours after symptom onset)
* Patients were able to complete cardiac magnetic resonance imaging (CMR) and speckle tracking imaging echocardiogram (STE) examinations
* Patients agreed and provided informed consent

Exclusion Criteria:

* Previous myocardial infarction or revascularization (PCI or CABG)
* Congestive heart failure with LVEF<40%
* Atrial fibrillation
* Renal insufficiency (GFR < 30 ml/min/1.73m^2)
* Acute infectious diseases within nearly 3 months
* Rheumatic immune system diseases
* Malignant tumors
* Claustrophobia
* Contraindicated to CMR
* Patients do not agree to be included in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to Beijing Friendship Hospital,Capital Medical University with a confirmed STEMI diagnosis undergoing primary percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
MACE (major adverse cardiovascular events) | 12 months
  nonfatal or fatal myocardial infarction, revascularization, cardiac death, nonfatal or fatal stroke, all cause of death

SECONDARY OUTCOMES:
adverse cardiac remodeling | 6 months
  a cut-off value of 12% change in left ventricular end-diastolic volume between the acute and follow-up magnetic resonance scans

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang Y, Gao H, Liu L, Li S, Hua B, Lan D, He Y, Li J, Chen H, Li W, Li H. Regulatory T Cell as Predictor of Intramyocardial Hemorrhage in STEMI Patients after Primary PCI. Rev Cardiovasc Med. 2023 Jul 14;24(7):205. doi: 10.31083/j.rcm2407205. eCollection 2023 Jul. PMID 39077002